CLINICAL TRIAL: NCT03151382
Title: A Based on PEEG and PET Study of Anxiolytic Treatment to Improve Cognitive Function in Patients With Alzheimer Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Enyan Yu, Secretary of Party Committee, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SED-AD; SED-AD-2016-001 (Other: Sumitomo Pharma （Suzhou） Co..Ltd)
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer Disease; Cognitive Function
Keywords: Alzheimer Disease; Cognitive Function; tandospirone
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Tandospirone Citrate; Drug: Donepezil Hydrochloride
- Control group (Other)
  Interventions: Drug: Donepezil Hydrochloride

INTERVENTIONS:
Drug: Tandospirone Citrate — Tandospirone, 30-60 mg/d
  Arms: Experimental group
Drug: Donepezil Hydrochloride — Donepezil, 10 mg/d

SUMMARY:
Objective: Evaluation the improvement of the cognitive function of tandospirone add-on treatment on patients with AD comorbid anxiety.

Number of Patients: 30

Methodology: Randomized, open-label, parallel-group

Assigned Interventions: Experimental: Tandospirone, 30-60 mg/d + Donepezil, 10 mg/d; Control group: Donepezil, 10 mg/d.

Effect Evaluation: Primary Outcome: Change from baseline in ADAS-cog total score at week 12; NPI scale total score at week 12;

ELIGIBILITY:
Inclusion Criteria:

* 55-80 years old (including 55 and 80), male or female, sufficient vision, hearing and general health to complete the follow-up and assessment;
* Patients who were diagnosed with AD according to the DSM-IV;
* MMSE score > 10 and ≤ 24;
* HAMA score > 8;
* HAMD score ≤ 7;
* Brain CT or MRI supports the diagnosis of AD;
* Provide written informed consent by the patient himself and his family member or guardian.

Exclusion Criteria:

* Dementia from any other cause;
* Brain MRI showed that the diameter of hyperintense lesions in T2-FLAIR sequences were larger than 5mm;
* Patients with significant cardiac, pulmonary, hepatic, renal, or hematologic disease;
* Any primary neurologic or psychiatric disease other than AD;
* Mental disorders due to substance abuse;
* Participation in other clinical studies within the last 30 days;
* History of alcohol or substance abuse or dependence within the past year;
* Pregnant or breastfeeding, or of child-bearing potential during the study.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-20 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of ADAS-cog total score | week 12
  Change from baseline in ADAS-cog total score at week 12
NPI scale total score | week 12
  NPI scale total score at week 12

SECONDARY OUTCOMES:
HAMA total score | week 12
  HAMA total score at week 12
FAB score | week 12
  FAB score at week 12
relative power | week 12
  Change from baseline in the relative power at week 12
the image of PET | week 12
  the image of PET at week 12
MMSE score | week 12
  MMSE score at week 12